CLINICAL TRIAL: NCT03392870
Title: Evaluation of a Clinical Program Specialized in the Diagnosis, Follow-up and Treatment of Young Adults With a Autism Spectrum Disorder: "TAVA" (Spanish Acronym for "Support to Subjects With Autism in Their Transition to Adulthood")
Brief Title: Evaluation of a Clinical Transitional Program in Autism
Acronym: TAVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Esther Via, Principal Investigator, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSPT04_TAVA
Record Dates: First submitted 2017-03-31; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Autism Spectrum Disorder (ASD); Transition program
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A researcher will be masked for group aleatorization (active, group) in order to unbiasedly evaluate outcomes which require subjective assesment of functionality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAVA-ACTIVE (Experimental): Integrative interventional programme. It involves high-frequency multidisciplinary intervention: nursing, psychology, psychiatry and social services. A psychotherapeutic group would be offered to those patients with an intelligence quotient>70, verbal communication and no behavioural alterations.
  Interventions: Other: Integrative interventional programme
- CONTROL (Active Comparator): As usual
  Interventions: Other: As usual

INTERVENTIONS:
Other: Integrative interventional programme — The active condition includes specialized, multidisciplinary and intensive individual (weekly to monthly) or group interventions (weekly). Only high-functioning subjects will be considered for group interventions.
  Arms: TAVA-ACTIVE
Other: As usual — The control group will follow treatment as usual, consisting in conventional general psychiatrist/psychologist clinical follow-up. The frequency varies between 3-6 months or 15-21 days if worsening of symptoms or comorbid conditions.
  Arms: CONTROL

SUMMARY:
Clinical trial without drug, randomized: Comparison of a specific and integrative clinical protocol for young adults with autism to usual treatment. It will include both low and high-functioning participants.

ELIGIBILITY:
Inclusion Criteria:

* ASD diagnosis
* Previous follow-up by child and adolescent psychiatry department at Corporació Sanitària Parc Taulí (CSPT)

Exclusion Criteria:

- Living in a disabled residential setting

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of life. | Baseline, 24 months
  The World Health Organization Quality of Life (WHOQOL). Self-administered scale, quantitative. Spanish version.

SECONDARY OUTCOMES:
Change in: Asperger Symptoms. | Baseline, 24 months
  Adult Asperger Assessment (AAA). Includes questionnaire (autism spectrum quotient, AQ) and (empathy quotient, EQ). Self-administered scale, quantitative.Spanish version.
Change in: Depressive symptoms | Baseline, 24 months
  Beck Depression Inventory-II (BDI-II) . Self-administered scale, quantitative.Spanish version.
Change in: Anxiety Symptoms. | Baseline, 24 months
  Beck Anxiety Inventory (BAI). Self-administered scale, quantitative.Spanish version.
Change in: Obsessive-compulsive symptoms. | Baseline, 24 months
  Obsessive-Compulsive Inventory - Revised (OCI-R). Self-administered scale, quantitative. Spanish version.
Change in: ASD symptoms evaluated by parents/caregiver. | Baseline, 24 months
  Social Responsiveness Scale (SRS). Parents' self-administered scale, quantitative.Spanish version.
Change in: ASD symptoms. | Baseline, 24 months
  Ritvo Autism Asperger's Diagnostic Scale (RAADS-R). Self-administered scale, quantitative. Spanish- translated version.
Change in: Social phobia symptoms. | Baseline, 24 months
  Social Phobia Inventory (SPIN). Self-administered scale, quantitative. Spanish version.
Change in: Evaluation of support needs. | Baseline, 24 months
  Camberwell Assessment of Need, revised (CAN-R). Administered by the professional, qualitative. Spanish version.
Change in: Caregiver's burden associated with the disorder. | Baseline, 24 months
  The Zarit Burden Interview. Caregiver self-report, quantitative. Spanish version.
Change in: Evaluation of the level of autonomy, self-regulation, self-empowerment, self-knowledge. | Baseline, 24 months
  The Arc's Self-Determination Scale. Self-administered scale. Spanish version. Quantitative.

CONTACTS AND LOCATIONS:
Overall Officials: ESTHER VIA, PHD, Principal Investigator — CORPORACIO SANITARIA PARC TAULI
Locations (1):
- Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No